CLINICAL TRIAL: NCT06050044
Title: Intrathecal Injection of Hyperbaric Bupivacaine Versus a Mixture of Hyperbaric and Isobaric Bupivacaine in Patients Undergoing Lower Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Intrathecal Injection of Hyperbaric Bupivacaine Versus a Mixture of Hyperbaric and Isobaric Bupivacaine in Patients Undergoing Lower Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Adel Ali Hassan, Lecturer of Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine, Helwan University, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48-2022
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Spinal Anesthesia; Hyperbaric Bupivacaine; Isobaric Bupivacaine; Lower Abdominal Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (hyperbaric bupivacaine) (Experimental): Patients were injected intrathecally with 20 mg hyperbaric bupivacaine 0.5% solution.
  Interventions: Drug: Group A (hyperbaric bupivacaine)
- Group B (Mixture of Hyperbaric and Isobaric Bupivacaine) (Experimental): Patients received 10 mg hyperbaric bupivacaine and 10 mg isobaric bupivacaine 0,5 % solution.
  Interventions: Drug: Group B (Mixture of Hyperbaric and Isobaric Bupivacaine)

INTERVENTIONS:
Drug: Group A (hyperbaric bupivacaine) — Patients were injected intrathecally with 20 mg hyperbaric bupivacaine 0.5% solution
  Arms: Group A (hyperbaric bupivacaine)
Drug: Group B (Mixture of Hyperbaric and Isobaric Bupivacaine) — Patients received 10 mg hyperbaric bupivacaine and 10 mg isobaric bupivacaine 0,5 % solution
  Arms: Group B (Mixture of Hyperbaric and Isobaric Bupivacaine)

SUMMARY:
The aim of this study is to compare the effects of intrathecal injection of hyperbaric bupivacaine versus injection of hyperbaric and isobaric bupivacaine in patients undergoing lower abdominal surgery.

DETAILED DESCRIPTION:
Spinal anesthesia is one of the most commonly used nerve block procedures for surgical operations involving the lower abdomen, the perineum, and the lower limbs, owing to its quick effect and cost-effectiveness. Spinal anesthesia is advantageous in that it uses a small dose of anesthesia, is simple to perform, and offers a rapid onset of action, reliable surgical analgesia, and good muscle relaxation.

The Baricity of a solution is defined as the ratio of the density of the solution to that of the cerebrospinal fluid (CSF). The most common anesthetic used for SA in obstetric and non-obstetric surgery is bupivacaine, which can be formulated as an isobaric or hyperbaric solution. Baricity differences between spinal anesthetic solutions are thought to affect hemodynamic parameters and distribution within the subarachnoid space, which may, in turn, affect the onset, extent, and duration of sensory block as well as side effects.

Spinal anesthesia has been linked to different adverse effects, out of which hypotension is most common complication. The incidence of hypotension is 25-75% in general population. Factors that increase the risk of hypotension include patient factors (advanced age, pregnancy, obesity, diabetes mellitus, hypertension, and anemia) and technical factors such as a block level at or above T5, use of opioids during premedication, and high local anesthetic dosages.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years old.
* Both sexes.
* American Society of Anaesthesia (ASA) I to II.
* Undergoing lower abdominal or urological surgery under spinal anesthesia

Exclusion Criteria:

* Allergy to amide.
* Patients with a significant history of substance abuse.
* Patients with diabetes mellitus, neurological or cardiovascular diseases.
* Patients with neuromuscular diseases.
* Pregnant patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | 3 hours post-injection
  Blood pressure was recorded using standard non-invasive monitors at 5, 10, 15, 20, 25, 30, 45, and 60 min, then hourly until 3 h post-injection.
  Hypotension was defined as a decrease in mean arterial pressure of more than 30% from baseline.

SECONDARY OUTCOMES:
Heart rate | 3 hours post-injection
  Heart rate was recorded using standard non-invasive monitors at 5, 10, 15, 20, 25, 30, 45, and 60 min, then hourly until 3 h post-injection.
Mean arterial pressure (MAP) | 3 hours post-injection
  Mean arterial pressure was recorded using standard non-invasive monitors at 5, 10, 15, 20, 25, 30, 45, and 60 min, then hourly until 3 h post-injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.